CLINICAL TRIAL: NCT05311410
Title: Viral Kinetics of SARS-CoV-2 in Patients in the Intensive Care Unit Undergoing Dental Procedures
Brief Title: Viral Kinetics of SARS-CoV-2 in Patients With COVID-19 in the Intensive Care Unit Undergoing Dental Procedures
Acronym: VKSPCICUDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Itamara Lucia Itagiba Neves, itamara@incor.usp.br, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-Dentistry
Record Dates: First submitted 2021-12-15; First posted 2022-04-05 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: SARS-CoV2 Infection; Viral Load; Oral Diseases; Dental Treatment
Keywords: COVID-19; Viral load; Dental treatment; Intensive care unit
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Non-bloody dental procedures (control group)
- Study group (Active Comparator)
  Interventions: Procedure: Bloody dental procedures (study group)

INTERVENTIONS:
Other: Non-bloody dental procedures (control group) — Control group composed of 30 positive patients for SARS-CoV-2, from the same ICU, submitted to non-bloody procedures.
  Arms: Control group
Procedure: Bloody dental procedures (study group) — Study group consisting of 30 patients who require open dental treatment and with a positive PCR test for SARS-CoV-2 prior and admitted to the Intensive Care Unit.
  Arms: Study group

SUMMARY:
The prevalence and clinical relevance of viremia in patients with COVID-19 have not been well investigated. Seeking to understand the need for dentistry to perform bloody procedures in critically ill patients with COVID-19 admitted to the ICU, the quantification of the magnitude of viral replication may play a fundamental role in this scenario. For this, it is necessary to study the viremia kinetics of SARS-CoV-2, seeking to assess whether there is any characteristic pattern that may be associated with a worse clinical outcome of the patient with COVID-19 after undergoing bloody dental procedures, therefore, the objective of this research will be to investigate the occurrence of viral kinetics produced by dental procedures in patients with SARS-CoV-2 in Intensive Care Units, where, in addition to analyzing the oral health condition, the viral kinetics of SARS-CoV-2 will also be investigated by means of reverse transcription polymerase chain reaction (RT-PCR) examination of blood samples from patients with COVID-19 undergoing bloody dental treatment. This research is expected to identify risks and consequences regarding the possibility of performing bloody dental treatment in patients with COVID-19 in serious condition, in addition to verifying the association of the impact of oral infection foci on this profile of patients.

ELIGIBILITY:
Inclusion Criteria: Patients between 16 and 90 years old who describe subgingival scaling of at least one dental sextant or a tooth extraction.

Exclusion Criteria: Patients who cannot perform clinical examination and/or open dental procedure.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Increased quantification of viral replication | Through three collections of blood samples, in the following moments: (T0) 15 minutes before the beginning of the dental procedure; (T1) 10 minutes after the start of the procedure; and (T3) 10 minutes after the end of the procedure.
  The performance of bloody dental procedures hospitalized critically ill patients with COVID-19 causes an increase in the quantification of viral replication, causing changes in the patient's clinical outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry Unit, Heart Institute, Clinical Hospital of the Faculty of Medicine of the University of São Paulo., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After the defense of the thesis, the digital file available on the Portal Digital Library of Theses and Dissertations of the University of São Paulo, in portable document format (PDF) file.

REFERENCES:
- [Background] Clerkin KJ, Fried JA, Raikhelkar J, Sayer G, Griffin JM, Masoumi A, Jain SS, Burkhoff D, Kumaraiah D, Rabbani L, Schwartz A, Uriel N. COVID-19 and Cardiovascular Disease. Circulation. 2020 May 19;141(20):1648-1655. doi: 10.1161/CIRCULATIONAHA.120.046941. Epub 2020 Mar 21. PMID 32200663
- [Background] Lai CC, Liu YH, Wang CY, Wang YH, Hsueh SC, Yen MY, Ko WC, Hsueh PR. Asymptomatic carrier state, acute respiratory disease, and pneumonia due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): Facts and myths. J Microbiol Immunol Infect. 2020 Jun;53(3):404-412. doi: 10.1016/j.jmii.2020.02.012. Epub 2020 Mar 4. PMID 32173241
- [Background] Backer JA, Klinkenberg D, Wallinga J. Incubation period of 2019 novel coronavirus (2019-nCoV) infections among travellers from Wuhan, China, 20-28 January 2020. Euro Surveill. 2020 Feb;25(5):2000062. doi: 10.2807/1560-7917.ES.2020.25.5.2000062. PMID 32046819
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Kinross P, Suetens C, Dias JG, Alexakis L, Wijermans A, Colzani E, Monnet DL; European Centre for Disease Prevention and Control (ECDC) Public Health Emergency Team; ECDC Public Health Emergency Team. Rapidly increasing cumulative incidence of coronavirus disease (COVID-19) in the European Union/European Economic Area and the United Kingdom, 1 January to 15 March 2020. Euro Surveill. 2020 Mar;25(11):2000285. doi: 10.2807/1560-7917.ES.2020.25.11.2000285. Epub 2020 Mar 16. PMID 32186277
- [Background] CDC COVID-19 Response Team. Preliminary Estimates of the Prevalence of Selected Underlying Health Conditions Among Patients with Coronavirus Disease 2019 - United States, February 12-March 28, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):382-386. doi: 10.15585/mmwr.mm6913e2. PMID 32240123
- [Background] Nguyen H, Manolova G, Daskalopoulou C, Vitoratou S, Prince M, Prina AM. Prevalence of multimorbidity in community settings: A systematic review and meta-analysis of observational studies. J Comorb. 2019 Aug 22;9:2235042X19870934. doi: 10.1177/2235042X19870934. eCollection 2019 Jan-Dec. PMID 31489279
- [Background] Dietz W, Santos-Burgoa C. Obesity and its Implications for COVID-19 Mortality. Obesity (Silver Spring). 2020 Jun;28(6):1005. doi: 10.1002/oby.22818. Epub 2020 Apr 18. No abstract available. PMID 32237206
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Radzikowska U, Ding M, Tan G, Zhakparov D, Peng Y, Wawrzyniak P, Wang M, Li S, Morita H, Altunbulakli C, Reiger M, Neumann AU, Lunjani N, Traidl-Hoffmann C, Nadeau KC, O'Mahony L, Akdis C, Sokolowska M. Distribution of ACE2, CD147, CD26, and other SARS-CoV-2 associated molecules in tissues and immune cells in health and in asthma, COPD, obesity, hypertension, and COVID-19 risk factors. Allergy. 2020 Nov;75(11):2829-2845. doi: 10.1111/all.14429. Epub 2020 Aug 24. PMID 32496587
- [Background] Amorim Dos Santos J, Normando AGC, Carvalho da Silva RL, Acevedo AC, De Luca Canto G, Sugaya N, Santos-Silva AR, Guerra ENS. Oral Manifestations in Patients with COVID-19: A Living Systematic Review. J Dent Res. 2021 Feb;100(2):141-154. doi: 10.1177/0022034520957289. Epub 2020 Sep 11. PMID 32914677
- [Background] Ahmed QA, Niederman MS. Respiratory infection in the chronically critically ill patient. Ventilator-associated pneumonia and tracheobronchitis. Clin Chest Med. 2001 Mar;22(1):71-85. doi: 10.1016/s0272-5231(05)70026-5. PMID 11315460
- [Background] Paju S, Scannapieco FA. Oral biofilms, periodontitis, and pulmonary infections. Oral Dis. 2007 Nov;13(6):508-12. doi: 10.1111/j.1601-0825.2007.01410a.x. PMID 17944664
- [Background] Marouf N, Cai W, Said KN, Daas H, Diab H, Chinta VR, Hssain AA, Nicolau B, Sanz M, Tamimi F. Association between periodontitis and severity of COVID-19 infection: A case-control study. J Clin Periodontol. 2021 Apr;48(4):483-491. doi: 10.1111/jcpe.13435. Epub 2021 Feb 15. PMID 33527378
- [Background] Holmgren CJ. CPITN--interpretations and limitations. Int Dent J. 1994 Oct;44(5 Suppl 1):533-46. PMID 7836008
- [Background] Chen L, Wang G, Long X, Hou H, Wei J, Cao Y, Tan J, Liu W, Huang L, Meng F, Huang L, Wang N, Zhao J, Huang G, Sun Z, Wang W, Zhou J. Dynamics of Blood Viral Load Is Strongly Associated with Clinical Outcomes in Coronavirus Disease 2019 (COVID-19) Patients: A Prospective Cohort Study. J Mol Diagn. 2021 Jan;23(1):10-18. doi: 10.1016/j.jmoldx.2020.10.007. Epub 2020 Oct 26. PMID 33122141
- [Background] Moreira MS, Neves ILI, de Bernoche CYSM, Sarra G, Dos Santos-Paul MA, Campos Neves da Silva F, Schroter GT, Montano TCP, de Carvalho CMA, Neves RS. Bilateral paresthesia associated with cardiovascular disease and COVID-19. Oral Dis. 2022 Apr;28 Suppl 1(Suppl 1):912-915. doi: 10.1111/odi.13539. Epub 2020 Aug 1. No abstract available. PMID 32640483
- [Background] Natoli S, Oliveira V, Calabresi P, Maia LF, Pisani A. Does SARS-Cov-2 invade the brain? Translational lessons from animal models. Eur J Neurol. 2020 Sep;27(9):1764-1773. doi: 10.1111/ene.14277. Epub 2020 May 22. PMID 32333487
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Corman VM, Landt O, Kaiser M, Molenkamp R, Meijer A, Chu DK, Bleicker T, Brunink S, Schneider J, Schmidt ML, Mulders DG, Haagmans BL, van der Veer B, van den Brink S, Wijsman L, Goderski G, Romette JL, Ellis J, Zambon M, Peiris M, Goossens H, Reusken C, Koopmans MP, Drosten C. Detection of 2019 novel coronavirus (2019-nCoV) by real-time RT-PCR. Euro Surveill. 2020 Jan;25(3):2000045. doi: 10.2807/1560-7917.ES.2020.25.3.2000045. PMID 31992387